CLINICAL TRIAL: NCT07032571
Title: Enhancing Weight Loss in a Digital Intervention Among Adults With Overweight or Obesity
Brief Title: Reset: Enhancing Weight Loss in a Digital Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Stanford Nutrition and Obesity Research Center (Unknown)
Responsible Party: Principal Investigator, Michele Patel, Principal Investigator, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 81144
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Overweight; Weight Loss; Health Behavior; Lifestyle Intervention
Keywords: obesity; overweight; weight loss; weight; health behavior; lifestyle intervention; lifestyle modification; multiphase optimization strategy; intervention; behavior change; weight reduction; lose weight; adults; BMI reduction; body fat reduction; weight control; weight change; weight management; obesity management; obesity treatment; digital health; digital intervention; remote intervention; standalone intervention; obesity prevention; diabetes prevention; mobile health; factorial design; intervention optimization
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Health Behavior; Body Weight; Body Weight Changes

STUDY DESIGN:
Intervention Model Description: This study uses a full factorial experimental design to test the impact of four intervention components, each with two levels, on vs. off (i.e., a 2x2x2x2, or 2^4 factorial design).
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be analyzed in a blinded fashion such that treatment allocation is not revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): Core Only
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention
- Condition 2 (Experimental): Core + Increase Fiber
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Increase Fiber Intake
- Condition 3 (Experimental): Core + Increase Protein
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Increase Protein
- Condition 4 (Experimental): Core + Increase Protein + Increase Fiber
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Increase Protein; Behavioral: Increase Fiber Intake
- Condition 5 (Experimental): Core + Limit Eating Window
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Eating Window
- Condition 6 (Experimental): Core + Limit Eating Window + Increase Fiber
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Eating Window; Behavioral: Increase Fiber Intake
- Condition 7 (Experimental): Core + Limit Eating Window + Increase Protein
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Eating Window; Behavioral: Increase Protein
- Condition 8 (Experimental): Core + Limit Eating Window + Increase Protein + Increase Fiber
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Eating Window; Behavioral: Increase Protein; Behavioral: Increase Fiber Intake
- Condition 9 (Experimental): Core + Limit Red Zone Foods
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Red Zone Foods
- Condition 10 (Experimental): Core + Limit Red Zone Foods + Increase Fiber
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Red Zone Foods; Behavioral: Increase Fiber Intake
- Condition 11 (Experimental): Core + Limit Red Zone Foods + Increase Protein
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Red Zone Foods; Behavioral: Increase Protein
- Condition 12 (Experimental): Core + Limit Red Zone Foods + Increase Protein + Increase Fiber
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Red Zone Foods; Behavioral: Increase Protein; Behavioral: Increase Fiber Intake
- Condition 13 (Experimental): Core + Limit Red Zone Foods + Limit Eating Window
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Red Zone Foods; Behavioral: Limit Eating Window
- Condition 14 (Experimental): Core + Limit Red Zone Foods + Limit Eating Window + Increase Fiber
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Red Zone Foods; Behavioral: Limit Eating Window; Behavioral: Increase Fiber Intake
- Condition 15 (Experimental): Core + Limit Red Zone Foods + Limit Eating Window + Increase Protein
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Red Zone Foods; Behavioral: Limit Eating Window; Behavioral: Increase Protein
- Condition 16 (Experimental): Core + Limit Red Zone Foods + Limit Eating Window + Increase Protein + Increase Fiber
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Limit Red Zone Foods; Behavioral: Limit Eating Window; Behavioral: Increase Protein; Behavioral: Increase Fiber Intake

INTERVENTIONS:
Behavioral: Core Behavioral Weight Loss Intervention — All participants receive a 12-week core behavioral weight loss intervention consisting of the following: daily self-monitoring of weight; weekly behavioral lessons and action plans to promote healthy eating and physical activity; and tailored feedback. The intervention will be delivered remotely via email and/or text message.
Behavioral: Limit Red Zone Foods — Participants randomized to receive this component are given a goal to limit their Red Zone Foods (i.e., foods high in calories and low in nutrition) and are instructed to self-monitor them daily.
  Arms: Condition 10; Condition 11; Condition 12; Condition 13; Condition 14; Condition 15; Condition 16; Condition 9
Behavioral: Limit Eating Window — Participants randomized to receive this component are given a goal to limit their eating windows (i.e., follow time-restricted eating) and are instructed to self-monitor them daily.
  Arms: Condition 13; Condition 14; Condition 15; Condition 16; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Increase Protein — Participants randomized to receive this component are given a goal to increase their protein intake and are instructed to self-monitor it daily.
  Arms: Condition 11; Condition 12; Condition 15; Condition 16; Condition 3; Condition 4; Condition 7; Condition 8
Behavioral: Increase Fiber Intake — Participants randomized to receive this component are given a goal to increase their fiber intake and are instructed to self-monitor it daily.
  Arms: Condition 10; Condition 12; Condition 14; Condition 16; Condition 2; Condition 4; Condition 6; Condition 8

SUMMARY:
The goal of the Reset trial is to learn about the optimal combination of dietary behavior strategies in a fully digital weight loss intervention. The intervention is designed for adults with overweight or obesity. The investigators will examine the impact on weight loss of four dietary strategies: 1) limiting Red Zone Foods (i.e., foods that are high in calories and low in nutrition), 2) limiting eating windows, 3) increasing protein intake, and 4) increasing fiber intake. Each of these strategies will include goal setting, daily self-monitoring, and tailored feedback.

The investigators will recruit 208 participants. Broadly, adults with overweight or obesity who live in the U.S. will be eligible. The weight loss intervention will last 12 weeks. All participants will be asked to track their body weight daily and complete weekly behavioral lessons and action plans to promote healthy eating and physical activity. All study tasks will occur remotely. Assessment of body weight and survey measures will occur at the beginning of the trial ("baseline"), and at 1 month and 3 months.

The Multiphase Optimization Strategy (MOST) framework will be used to identify which combination of the dietary behavior strategies results in the greatest weight loss. In total, there will be 16 treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* adults (ages 18+ years)
* body mass index (BMI) 25.0 to 45.0 kg/m^2
* cellphone ownership with a texting plan
* daily access to a personal scale
* daily access to a personal email account
* English language proficiency
* interest in losing weight through behavioral strategies
* living in the United States

Exclusion Criteria:

* concurrent enrollment in another weight management intervention
* loss of ≥5% body weight in the past 6 months
* current use of a weight loss or anti-obesity medication
* prior or planned bariatric surgery in the next 3 months
* current pregnancy, planned pregnancy in the next 3 months, or recent pregnancy in the past 6 months
* current breastfeeding or lactating
* living with someone else participating in the study
* hospitalization for a mental health condition in the past 12 months
* inability to engage in moderate forms of physical activity akin to brisk walking
* if weight loss is contraindicated or might be impacted by a condition (e.g., end stage renal disease, cancer, schizophrenia, dementia) or medication (e.g., steroids, antipsychotics)
* if an individual would be better suited for a more intensive or different type of intervention based on a health condition (e.g., individuals with history of an eating disorder or cardiovascular event, uncontrolled hypertension, or uncontrolled diabetes mellitus)
* participation in another weight loss study conducted in Dr. Patel's lab in the past 6 months
* investigator discretion for safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Weight Change from Baseline to 3 Months | Baseline and 3 Months
  mean change in kg; assessed via participants' personal scales

SECONDARY OUTCOMES:
Weight Change from Baseline to 1 Month | Baseline and 1 Month
  mean change in kg; assessed via participants' personal scales
Clinically Significant Weight Loss at 3 Months | 3 Months
  operationalized as the proportion of participants achieving ≥5% weight loss from baseline
Moderate-to-Vigorous Physical Activity (MVPA) Change from Baseline to 3 Months | Baseline and 3 Months
  mean change; assessed via the Godin Leisure-Time Exercise Questionnaire (GLTEQ)'s MVPA Score Index. The GLTEQ is a self-report measure that assesses a typical week's frequency of engaging in different types of exercise (strenuous, moderate, mild/light) for at least 15 minutes. Minimum score is 0. Higher scores indicate more frequent exercise. Scores ≥ 24 indicate "active" while scores < 24 indicate "insufficiently active."
Caloric Intake Change from Baseline to 3 Months | Baseline and 3 Months
  mean change in kilocalories; assessed via the Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24): 2 separate 24-hour diet recalls per time point: 1 week day, 1 weekend day

OTHER OUTCOMES:
Engagement in Self-Monitoring Weight | Weeks 1 to 12
  operationalized as average percentage of days in the 12-week intervention with self-monitoring of weight; assessed via scale (then logged via text message or daily e-checklist); will report median (IQR) if non-normally distributed
Engagement in Self-Monitoring Eating Behaviors | Weeks 1 to 12
  operationalized as average percentage of days in the 12-week intervention with self-monitoring of eating behaviors; assessed via daily e-checklist; will report median (IQR) if non-normally distributed

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Patel, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified dataset and metadata will be made available through a public repository. It will include the primary outcome (weight change), secondary outcomes, and participant level characteristics. Data will be available in an Excel spreadsheet, whereby each row corresponds to a unique participant's data, and columns represent the different variables mentioned, by time point.
Supporting Information: Study Protocol, SAP
Time Frame: The shared dataset will be made publicly available upon publication of the primary outcomes in a peer-reviewed journal.
Access Criteria: Publicly available.